CLINICAL TRIAL: NCT07179978
Title: Lorazepam Dose and the Risk of Serious Adverse Events in Older Adults With Low Kidney Function: A Population-Based Cohort Study Research Protocol
Brief Title: Lorazepam and the Risk of Serious Adverse Events
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: 2025 0906 609 0001; ICES # 2025 0906 609 001 (Other: Canadian Institutes of Health Research)
Record Dates: First submitted 2025-09-05; First posted 2025-09-18 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Chronic Kidney Disease (CKD)
Keywords: chronic kidney disease; older adults; benzodiazepines; adverse events; cohort study; drug safety; lorazepam; sleeping pills; gediatrics
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Lorazepam

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High dose of lorazepam (>1-4 mg/day): Residents of Alberta and Ontario, aged 66 years or older with low kidney function (an eGFR <45 mL/min per 1.73 m2 but not receiving dialysis or having a history of kidney transplantation) who have filled a new oral prescription for lorazepam (high-dose >1-4 mg/day) at an outpatient pharmacy under the Ontario Drug Benefit (ODB) program from January 01, 2008, to September 1, 2024, with a day supply of ≥5 days. The date when the prescription was filled will serve as the patient's entry or index date for the cohort, and each patient will enter the cohort only once. The accrual period for Alberta will be determined.
  Interventions: Drug: Lorazepam
- Low-dose of lorazepam (0.5-1 mg/day): Residents of Ontario and Alberta, aged 66 years or older with low kidney function (an eGFR <45 mL/min per 1.73 m2 but not receiving dialysis or having a history of kidney transplantation) who have filled a new oral prescription for lorazepam (low-dose 0.5-1 mg/day) at an outpatient pharmacy under the Ontario Drug Benefit (ODB) program from January 01, 2008, to September 1, 2024, with a day supply of ≥5 days. The date when the prescription was filled will serve as the patient's entry or index date for the cohort, and each patient will enter the cohort only once. The accrual period for Alberta will be determined.
  Interventions: Drug: Lorazepam

INTERVENTIONS:
Drug: Lorazepam — The primary exposure of interest will be oral lorazepam at a dose range of >1-4 mg/day.

SUMMARY:
This is a population-based cohort study assessing whether initiating a new outpatient prescription of a higher dose of lorazepam (>1-4 mg/day) compared to a lower dose (0.5-1 mg/day) in older adults with low kidney function (an eGFR <45 mL/min per 1.73 m2 but not receiving dialysis or having a history of kidney transplantation) is associated with an increased 30-day risk of a composite outcome, including all-cause hospitalization, all-cause emergency visit, or all-cause mortality.

DETAILED DESCRIPTION:
*Summary*

Background:

Benzodiazepine use in older adults is associated with a higher risk of falls, fractures, hospitalizations, emergency visits, and mortality. Despite warnings from Health Canada against prescribing benzodiazepines to older adults, approximately 1 in 9 adults aged 65+ were prescribed a benzodiazepine in 2019 in Ontario. Lorazepam is a commonly prescribed benzodiazepine for the management of insomnia and anxiety. It is primarily excreted in the urine. In patients with low kidney function, especially older adults, lorazepam can accumulate and increase the risk of developing serious adverse events.

The most common measure to assess kidney function in routine clinical care is the estimated glomerular filtration rate (eGFR), expressed in lab reports as mL/min/1.73 m2. A normal eGFR is >90 mL/min/1.73 m2, and a value <45 mL/min/1.73 m2 is considered to be low.

Prescribing references, product monographs, and other standard sources do not provide lorazepam daily dose recommendations in patients with low kidney function. As a result, lorazepam is often initiated at the standard doses in patients with low kidney function.

The investigators aim to conduct a population-based cohort study among older adults with low kidney function in two Canadian provinces, Alberta and Ontario, comparing the risk of serious adverse events among those initiating a higher dose versus a lower dose of lorazepam in the outpatient setting.

Methods: In this population-based retrospective cohort study, eligible participants will include older adults (≥66 years) with eGFR <45 mL/min/1.73 m2 (not receiving dialysis or having a history of kidney transplantation) from Alberta and Ontario who were dispensed a new outpatient prescription for oral lorazepam (0.5-4 mg/day) with a day supply of ≥5 days. In Ontario, accrual will occur between January 1, 2008, and September 1, 2024; the study period in Alberta will be determined based on data availability. Based on the prescribed daily dose, individuals will be divided into two groups: low-dose (0.5-1 mg/day) and high-dose (>1-4 mg/day). Propensity score weighting will be used to ensure both groups are well-balanced on a comprehensive set of measured baseline characteristics.

The primary outcome will be a 30-day composite of all-cause hospitalization, emergency department visit, and mortality.

*Background* Lorazepam is a commonly prescribed benzodiazepine used for the management of insomnia and anxiety in older adults with low kidney function.

Current lorazepam daily dose recommendations in this population are variable, ranging from 0.5 to 4 mg/day. Lorazepam use in older adults has been associated with a higher risk of serious adverse events, including falls, fractures, hospitalizations, emergency visits, and mortality.

Understanding the risks of initiating higher versus lower doses of lorazepam in older adults with low kidney function can be used to guide safe prescribing and better outcomes in this population.

*Objectives*

Is there a higher 30-day risk of a composite outcome of all-cause hospitalization, or all-cause emergency visit, or all-cause mortality among older adults with low kidney function (an eGFR <45 mL/min per 1.73 m2 but not receiving dialysis or having a history of kidney transplantation) who initiate a high dose (>1-4 mg/day) versus a low dose (0.5-1 mg/day) lorazepam in the outpatient setting?

*Study Design and Setting*

The investigators propose a population-based retrospective cohort study using linked administrative health data from Alberta and Ontario, Canada's two largest provinces.

Ontario data will be sourced from ICES (ices.on.ca). It offers secure, encrypted individual-level data for Ontario residents, all with universal access to hospital and physician services under a government-funded, single-payer healthcare system. The use of data in this study is authorized under section 45 of Ontario's Personal Health Information Protection Act, which does not require review by a research ethics board. The information needed for analyzing the primary outcomes is available across specific databases within the ICES system: data on all-cause hospitalizations are available in the Canadian Institute for Health Information Discharge Abstract Database, emergency visits in the National Ambulatory Care Reporting System, and mortality in the Registered Persons Database.

Alberta data will be accessed through the Alberta Kidney Disease Network. This dataset ends in ~ 2021.

The investigators are publicly registering our study protocol and documenting the study description, design, and statistical analysis prior to conducting outcome analyses. The results of this study will be reported adhering to RECORD reporting guidelines.

*Study Population*

The investigators will include all older adults (≥66 years) with an eGFR <45 mL/min per 1.73 m2 (not receiving dialysis or having a history of kidney transplantation) who received a new outpatient prescription for oral lorazepam with an initial dose between 0.5 and 4 mg/day and a day supply of ≥5 days. The dispensing date of the prescription will serve as the index date, and only the first eligible prescription will be included to ensure unique cohort entry, and each individual can enter the cohort only once.

*Baseline Characteristics*

Health records, census files, hospital discharge records, laboratory data, and physician claims will provide baseline variables, including demographic characteristics (such as age, sex, rurality, neighborhood income quintile), comorbidities, and medication use. Baseline comorbidities and healthcare utilization will be assessed using 5-year and 1-year look-back periods from the index date. Baseline medication use will be assessed within 120 days prior to the index date.

*Outcomes*

Participant observation time will be censored at the time of the first occurrence of the outcome of interest, death (if not the outcome of interest), or 30 days after the index date, whichever comes first.

The primary outcome is a 30-day composite outcome of all-cause hospitalization, all-cause emergency visit, and all-cause mortality.

Secondary outcomes will include

* Components of the primary composite outcome: 30-day all-cause hospitalization, all-cause emergency visit, and all-cause mortality, each examines separately.
* 30-day composite outcome of a hospital encounter (hospital admission or emergency visit) with delirium or encephalopathy (disorientation, transient alteration of awareness, other and unspecified symptoms and signs involving cognitive function) or hospital admission with receipt of an urgent computed tomography scan of the head.
* 30-day composite outcome of a hospital encounter (hospital admission or emergency visit) with fragility fracture (hip, femur, humerus, wrist/forearm, pelvis, and spine), falls, hypotension, or syncope

*Statistical analysis plan*

In Canada, the investigators are unable to connect individual-level patient data from different provinces due to privacy concerns. However, the investigators will combine results from both provinces (Alberta and Ontario) using the method outlined in a later section of this protocol.

Categorical variables will be summarized as frequencies and proportions, while continuous variables will be summarized as means with standard deviations (SD) or medians with interquartile ranges (IQR), as appropriate.

Baseline characteristics will be compared between the high-dose (>1-4 mg/day) and the low-dose (0.5-1 mg/day) groups using standardized mean differences (SMDs), with an absolute SMD greater than 10% considered indicative of a meaningful imbalance.

Balancing comparator group: The investigators will use inverse probability of treatment weighting (IPTW) on the propensity score to balance baseline characteristics between the high-dose (>1-4 mg/day) and low-dose (0.5-1 mg/day) groups, including known predictors of lorazepam use.

Propensity scores will be generated using a multivariable logistic regression model with all baseline characteristics.

Average treatment effect in the treated (ATT) weights will be used, where patients in the low-dose group will be assigned weights calculated as (propensity score / [1 - propensity score]) and patients in the high-dose group will receive a weight of 1. This method will produce a weighted pseudo-sample of patients in the referent group, i.e., low-dose lorazepam (0.5-1 mg/day), with a similar distribution of measured baseline characteristics as the high-dose lorazepam (>1-4 mg/day) group. Baseline characteristics will be compared between groups using standardized differences in both unweighted and weighted samples.

Regression analysis: To evaluate the primary outcome composite measure of all-cause hospitalization, all-cause emergency department visit, or all-cause mortality, the investigators will apply a modified Poisson regression analysis to estimate the risk ratio (95% CI) and binomial regression to estimate the risk difference (95% CI) using the weighted cohort, with the low-dose lorazepam (0.5-1 mg/day) group as the referent.

Secondary analyses:

The investigators will conduct independent testing for all secondary outcomes without adjusting for multiple comparisons. Each test will be performed and reported independently. In line with best practices, the primary outcome will be presented with its P-value, and the investigators will report all secondary outcomes using point estimates with 95% confidence intervals.

Additional analyses: The investigators plan to conduct four additional analyses.

1. Effect measure modification (EMM):

   For EMM, the investigators will expand our cohort to all the eGFR levels and categorize them into three groups: eGFR ≥60, 45-<60, and <45 mL/min/1.73 m2. Baseline characteristics between high-dose (>1-4 mg/day) and low-dose (0.5-1 mg/day) lorazepam groups will be assessed using standardized differences for all renal function categories combined and then within each of three eGFR categories (≥60, 45-<60, and <45 mL/min/1.73 m²).

   To further balance baseline characteristics between high-dose and low-dose lorazepam groups, the investigators will apply the IPTW method (described above), based on propensity scores for all the eGFR categories combined and within each of the three eGFR categories.

   EMM on the absolute scale for the primary composite outcome (30-day composite outcome of all-cause hospitalization, all-cause emergency visit, or all-cause mortality) will be examined across three baseline eGFR categories.

   EMM will be assessed on both the additive and multiplicative scales.
   * For additive interaction, the investigators will use binomial regression with an identity link to estimate risk differences, including an interaction term between low-dose and high-dose lorazepam groups and eGFR strata.
   * For multiplicative interaction, the investigators will use modified Poisson regression analysis to estimate risk ratios, including an interaction term between low-dose and high-dose lorazepam groups and eGFR strata.
2. Our interest in examining the safety of lorazepam in older adults with low kidney function is derived from high-throughput computing analysis in which the investigators executed 700+ population-based, new-user cohort studies, each comparing 74 acute (30-day) outcomes across strata of kidney function (PMID: 38186562). In this analysis, lorazepam was compared against non-users; the investigators found signs of harm, prompting us to undertake the current study. High-throughput analysis was run using Ontario data from January 1, 2008, to March 1, 2020. To confirm results, when there is no overlap, the investigators will run our analysis restricting the cohort after March 1, 2020.

   Examine whether the association between high-dose (>1-4 mg/day) versus low-dose (0.5-1 mg/day) lorazepam and the primary outcome is different (modified) in 2 period categories (the period before the end date of the high-throughput computing, and the period after the end date of the high-throughput computing).

   The investigators will perform analysis restricted to the non-overlap period, i.e., after March 1, 2020.
3. Compute the hazard ratio for all outcomes within 30 days, illustrating the effect of the intervention on each outcome over time. The investigators expect hazard ratios results similar to risk ratios. Although the difference between hazard ratios and risk ratios may be minimal over a short follow-up period, the hazard ratio offers additional insight by accounting for time-to-event analysis.
4. Perform E-value analyses to determine the minimum association strength an unmeasured confounder would need with both the prescription drug and the outcome of interest to eliminate the observed association.

*Combining Outcome Results from Alberta and Ontario* The investigators will use a privacy-preserving method to combine Alberta and Ontario's outcome results, while maintaining data privacy and regulatory compliance.

The investigators will use a privacy-preserving Cox-based approach for estimating risk ratios for multisite studies where individual-level data cannot be shared due to privacy constraints. The proposed method requires only a single transfer of summary-level outputs from each province to the research team. It produces results identical to those from the modified Poisson regression with combined individual-level data. The method was developed by adapting the risk-set table approach for survival outcomes, assuming stratified province-specific baseline risks, and allowing for confounding mitigation strategies such as propensity score matching or weighting to be done individually in each province. Each province will independently calculate these summary tables using their individual-level data. The summary-level risk-set tables generated in Alberta and Ontario will be shared with the research team, where they will be used to estimate the combined risk ratios and 95% confidence intervals. This will enable a robust and consistent analysis while maintaining data privacy and adhering to regulatory compliance. To comply with privacy regulations for minimizing the chance of identification of any individual, in all manuscripts, the number of individuals will be suppressed in the case of 5 or fewer participants (reported as ≤5).

ELIGIBILITY:
Inclusion Criteria:

The cohort will include older adults aged 66 years or greater with low kidney function (an eGFR <45 mL/min per 1.73 m2 but not receiving dialysis or having a history of kidney transplantation) who have filled a new oral prescription for lorazepam at an outpatient pharmacy with a dose range of 0.5-4 mg/day and a day supply of ≥5 days from January 1, 2008, to September 1, 2024 for Ontario; dates in Alberta to be finalized based on data availability.

Exclusion Criteria:

1. Individuals with missing administrative database number, missing or invalid age (<0 or >105 years), missing or invalid sex, death on or before the index date, non-Ontario resident (for Ontario data), or non-Alberta residents (for Alberta data).
2. Individuals less than 66 years of age on the index date.
3. Those with evidence of any study drug prescription 180 days before the index date (to restrict to new users only).
4. Individuals with other benzodiazepine and benzodiazepine-related drugs (alprazolam, bromazepam, chlordiazepoxide, clobazam, clonazepam, clorazepate, diazepam, ketazolam, midazolam, estazolam, flurazepam, nitrazepam, oxazepam, temazepam, triazolam, eszopiclone, zopiclone, and zolpidem) prescription in the previous 180 days before the index date or on the index date.
5. Individuals with more than one study drug prescription on the index date, as this complicates the ability to ascertain the prescribed dose accurately.
6. Evidence of other related drugs (melatonin, trazodone, doxepin, and suvorexant) and non-oral formulations of the study drugs in the previous 180 days, including the index date.
7. Individuals with end-stage renal disease, chronic dialysis, or a kidney transplant prior to the index date.
8. Evidence with hospital discharge or emergency department visit in the two days prior to or on the index date to ensure a new outpatient prescription.
9. Individuals with no serum creatinine lab value in the 0-365 days prior to the index date.
10. Individuals with unstable baseline kidney function:

    * If the most recent serum creatinine test prior to the index date was an inpatient test [ER or hospitalization] <refer to this as test date 1>, and there is not at least one 'outpatient' serum creatinine in the year before test date 1, OR
    * If the most recent prior serum creatinine test prior to the index date was an inpatient test [ER or hospitalization] <refer to this as test date 1>, and while there is at least 'outpatient' serum creatinine test in the year before <test date 1>, the most recent outpatient test prior to <test date 1> differs by an eGFR 10 mL/min/1.73 m2 or more from the value on <test date 1>.

    In Ontario, it has been shown that outpatient serum creatinine measurements in the province, conducted on a single occasion, indicate stable values.
11. Individuals receiving palliative care in the 0-365 days prior to the index date, in this setting, dosing is less relevant; rather, the focus is comfort care.

The investigators restrict to the first prescription in individuals with more than one eligible prescription. Date of this prescription will be the index date (the Date from which the outcomes start being assessed).

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Adults aged 66 years or older with low kidney function (eGFR <45 mL/min per 1.73 m2 but not receiving dialysis or having a history of kidney transplantation) who have filled a new outpatient prescription for lorazepam with a dose range of 0.5-4 mg/day and a day supply of ≥5 days between 2008 and 2024 in Ontario. The study accrual period for Alberta will be determined based on data availability.
Sampling Method: Non-Probability Sample
Enrollment: 12308 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with a composite outcome of all-cause hospitalization, all-cause emergency visit, or all-cause mortality. | Older adults exposed to high-dose (>1-4 mg/day) vs low-dose (0.5-1 mg/day) lorazepam will enter the cohort and will be followed until study outcome (first event), death, or 30 days from the cohort entry date.
  All-cause hospitalization, all-cause emergency visit, and all-cause mortality will be combined into a composite measure. Only the first hospitalization or emergency department visit occurring after the cohort entry date will be considered.

SECONDARY OUTCOMES:
Number of participants with all-cause hospitalization. | Older adults exposed to high-dose (>1-4 mg/day) vs low-dose (0.5-1 mg/day) lorazepam will enter the cohort and will be followed until study outcome (first event), death, or 30 days from the cohort entry date.
  One of the components of the primary composite outcome, all-cause hospitalization, individually presented as a secondary outcome. Only the first hospitalization after the cohort entry date will be considered.
Number of participants with all-cause emergency department visit. | Older adults exposed to high-dose (>1-4 mg/day) vs low-dose (0.5-1 mg/day) lorazepam will enter the cohort and will be followed until study outcome (first event), death, or 30 days from the cohort entry date.
  One of the components of the primary composite outcome, all-cause emergency department visit, individually presented as a secondary outcome. Only the first emergency department visit after the cohort entry date will be considered.
Number of participants with all-cause mortality | Older adults exposed to high-dose (>1-4 mg/d) vs low-dose (0.5-1 mg/d) lorazepam will enter the cohort and will be followed until study outcome (first event), death, or 30 days from the cohort entry date.
  One of the components of the primary composite outcome, all-cause mortality, individually presented as a secondary outcome.

OTHER OUTCOMES:
30-day composite outcome of a hospital encounter with delirium, encephalopathy, or hospital admission with receipt of an urgent computed tomography scan of the head | Older adults exposed to high-dose (>1-4 mg/day) vs low-dose (0.5-1 mg/day) lorazepam will enter the cohort and will be followed until study outcome (first event), death, or 30 days from the cohort entry date.
  30-day composite outcome of a hospital encounter (hospital admission or emergency visit) with delirium or encephalopathy (disorientation, transient alteration of awareness, other and unspecified symptoms and signs involving cognitive function) or hospital admission with receipt of an urgent computed tomography scan of the head.
30-day composite outcome of a hospital encounter with fragility fracture, falls, hypotension, or syncope. | Older adults exposed to high-dose (>1-4 mg/day) vs low-dose (0.5-1 mg/day) lorazepam will enter the cohort and will be followed until study outcome (first event), death, or 30 days from the cohort entry date.
  30-day composite outcome of a hospital encounter (hospital admission or emergency visit) with fragility fracture (hip, femur, humerus, wrist/forearm, pelvis, and spine), falls, hypotension, or syncope.

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre Research Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The dataset from this study is held securely in coded form at ICES. While legal data sharing agreements between ICES and data providers (e.g., healthcare organizations and government) prohibit ICES from making the dataset publicly available, access may be granted to those who meet pre-specified criteria for confidential access, available at www.ices.on.ca/DAS (email: das@ices.on.ca). The full dataset creation plan and underlying analytic code are available from the authors upon request, understanding that the computer programs may rely upon coding templates or macros that are unique to ICES and are therefore either inaccessible or may require modification.

REFERENCES:
- [Background] Shu D, Zou G, Hou L, Petrone AB, Maro JC, Fireman BH, Toh S, Connolly JG. A simple Cox approach to estimating risk ratios without sharing individual-level data in multisite studies. Am J Epidemiol. 2025 Jan 8;194(1):226-232. doi: 10.1093/aje/kwae188. PMID 38973755
- [Result] Abdullah SS, Rostamzadeh N, Muanda FT, McArthur E, Weir MA, Sontrop JM, Kim RB, Kamran S, Garg AX. High-Throughput Computing to Automate Population-Based Studies to Detect the 30-Day Risk of Adverse Outcomes After New Outpatient Medication Use in Older Adults with Chronic Kidney Disease: A Clinical Research Protocol. Can J Kidney Health Dis. 2024 Jan 6;11:20543581231221891. doi: 10.1177/20543581231221891. eCollection 2024. PMID 38186562